CLINICAL TRIAL: NCT07282301
Title: Evaluation of the Clinical Outcomes of the Embolic Protection System in Preventing Distal Embolism During Femoropopliteal Debulking Procedures
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); First Affiliated Hospital of Zhejiang University (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Huashan Hospital (Other); Shanghai Zhongshan Hospital (Other); Qingdao Haici Hospital (Other); Ruijin Hospital (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Chengdu University of Traditional Chinese Medicine (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Other Study IDs: the EPISODE study
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Femoropopliteal Disease
Keywords: Embolic Protection System; Distal embolism; Debulking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Embolic Protection System during femoropopliteal endovascular debulking: Using Embolic Protection System for preventing distal embolism during femoropopliteal endovascular debulking
  Interventions: Device: Embolic Protection System

INTERVENTIONS:
Device: Embolic Protection System — Using Embolic Protection System for preventing distal embolism during femoropopliteal endovascular debulking procedures

SUMMARY:
Patients with femoropopliteal arterial lesions requiring debulking procedures. The objective of this study is Evaluation of the clinical outcomes of the Embolic Protection System for preventing distal embolism during femoropopliteal endovascular debulking procedures (The EPISODE study).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Rutherford classification 2-5
3. Patients with chronic femoropopliteal obstruction or thromboembolism who require debulking prior to other endovascular treatments.
4. Patients who understand the purpose of this study, participate in the study voluntarily, sign the informed consent and are willing to receive follow-up visits
5. The guidewire needs to pass through the lesion
6. Life expectancy >24 months
7. Moderate to severe calcified lesions confirmed by imaging
8. For patients who receive intervention in both lower extremities, they may be enrolled in order of time of endovascular therapy
9. For combined aortoiliac artery lesions, recanalization of blood flow through endoluminal reconstruction of the vessel without more than 50% residual stenosis.

Exclusion Criteria:

1. Patients with stroke, cerebral hemorrhage, gastrointestinal hemorrhage, or cardiac infarction within 3 months prior to enrollment
2. Patients with known allergy to heparin, aspirin, other antiplatelet drugs, contrast agents, etc.
3. Patients who have been treated with drugs that interfere with this clinical trial or intraoperatively with other special vascular bed preparation devices, such as plaque volume reduction devices, special balloons, etc., within the last 3 months;
4. Pregnant and lactating women
5. Patients who are unable or unwilling to participate in this trial
6. patients with Berger's disease
7. Patients who have undergone arterial bypass on the treated side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients using Embolic Protection System for preventing distal embolism during femoropopliteal endovascular debulking procedures
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day freedom from Major adverse events (MAEs) | 30 days after intervention
  Incidence of no major adverse events within 30 days. Major adverse event is defined as death; acute cardiac infarction; unplanned amputation; acute thrombosis of the target vessel; serious complications related to the filter, such as vessel perforation, detachment of the filter, and severe entrapment (type D,E,F); distal embolism with clear clinical signs (specifically, the presence of imaging evidence of clear distal embolism at the distal end of the filter, with severe manifestations of ischemia that require further endoluminal or surgical intervention for relief, or cause tissue damage/longer hospitalization).

SECONDARY OUTCOMES:
Device Success Rate | Immediately after intervention
  Defined as: the filter passes through the lesion smoothly and is fully released distal to the lesion, and could be retrieved smoothly at the end of the treatment without serious vascular entrapment, distal embolization, or vascular perforation during release and retrieval
Technical success rate | Immediately after intervention
  Defined as: successful revascularization without termination of operation due to device

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No